CLINICAL TRIAL: NCT02342665
Title: Open-label, Uncontrolled, Single-arm, Phase Ib/II Study of Intravenous Copanlisib in Japanese Patients With Indolent B-cell Non Hodgkin's Lymphomas Relapsed After or Refractory to Standard Therapy
Brief Title: Japanese Phase Ib/II Copanlisib in Relapsed, Indolent B-cell NHL
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17792
Record Dates: First submitted 2015-01-15; First posted 2015-01-21 (Estimated); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Lymphoma Non-Hodgkin
Keywords: Non Hodgkin's Lymphomas
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — copanlisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Copanlisib (BAY80-6946) (Experimental): Dose escalation/safety evaluation cohort and objective tumor response (OR) expansion cohort
  Interventions: Drug: Copanlisib (BAY80-6946)

INTERVENTIONS:
Drug: Copanlisib (BAY80-6946) — Dosing is weekly for the first 3 weeks (on Days 1, 8, and 15) of a 28-day cycle, followed by a 1-week break (i.e., no infusion on Day 22).

SUMMARY:
The primary objective of this study is to assess the safety profile of copanlisib at the recommended dose (primary endpoint). The recommended dose of copanlisib for Japanese patients will be determined in the dose escalation/safety evaluation part.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of indolent B-cell NHL, with histological subtype limited to the following:

Follicular lymphoma (FL) grade 1-2-3a Small lymphocytic lymphoma (SLL) with absolute lymphocyte count < 5 x 109/L at the time of diagnosis and at study entry Lymphoplasmacytoid lymphoma/Waldenström macroglobulinemia (LPL/WM) Marginal zone lymphoma (MZL) (splenic, nodal, or extra-nodal)

* Relapsed or refractory after ≥ 2 prior lines of therapy (refractory defined as not responding to a standard regimen or progressing within 6 months of the last course of a standard regimen). Patients must have previously received rituximab and alkylating agent(s).
* Japanese patients ≥ 20 years of age
* ECOG performance status ≤ 2 (Eastern Cooperative Oncology Group:ECOG)
* Life expectancy of at least 3 months
* Adequate bone marrow, liver and renal function as assessed within 7 days before starting study treatment
* Left ventricular ejection fraction (LVEF) ≥ lower limit of normal (LLN) for the Institution
* Availability of fresh or archival tumor tissue

Exclusion Criteria:

* Uncontrolled hypertension (blood pressure ≥ 150/90 mmHg, defined as systolic blood pressure > 150 mmHg and/or diastolic blood pressure > 90 mmHg, despite optimal medical management)
* Patients with evidence or history of bleeding diathesis. Any hemorrhage or bleeding event ≥ CTCAE Grade 3 (NCI-CTC version 4.0) within 4 weeks of start of study medication (CTCAE: Common Terminology Criteria for Adverse Events, NCI: National Cancer Institute).
* History or concurrent condition of interstitial lung disease or severely impaired pulmonary function
* Unresolved toxicity higher than CTCAE grade 1 attributed to any prior therapy/procedure excluding alopecia.
* Prior treatment with PI3K inhibitors
* Systemic corticosteroid therapy (ongoing)
* Type I or II diabetes mellitus with HbA1c > 8.5% or fasting plasma glucose > 160 mg/dL at Screening
* Known history of human immunodeficiency virus (HIV) infection.
* Hepatitis B or C requiring treatment
* Cytomegalovirus (CMV) PCR positive at baseline
* Known lymphomatous involvement of the central nervous system

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | Up to 18 months
Intensity of AE | Up to 18 months
  The NCI Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0) will be used to assess the intensity of AE
Objective Tumor Response (OR) | Up to 18 Years
  OR: Best response rating of complete response or partial response according to the criteria defined in the Revised Response Criteria for Malignant Lymphoma(JClin Oncol.2007 Feb)
Recommended dose determined in the dose escalation/safety evaluation | Up to 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (8):
- Japan (8):
  - Nagoya, Aichi-ken
  - Maebashi, Gunma
  - Kobe, Hyōgo
  - Sendai, Miyagi
  - Chuo-ku, Tokyo
  - Koto-ku, Tokyo
  - Fukuoka
  - Kyoto

REFERENCES:
- See also: Click here to find information for studies related to Bayer products. To find this study enter the ClinicalTrials.gov identifier (NCT) number or Bayer Study Identifier (ID) in the search field. — http://clinicaltrials.bayer.com/